CLINICAL TRIAL: NCT01789268
Title: Impact of Respiratory Virus Infections and Bacterial Microbiome Shifts on Lymphocyte and Respiratory Function in Infants Born Prematurely or Full Term
Brief Title: Impact of Respiratory Pathogens in Infants
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Gloria Pryhuber, Professor, University of Rochester
Other Study IDs: 12-0012; 272201200005C-P00025-9999-5 (NIH)
Record Dates: First submitted 2013-02-07; First posted 2013-02-12 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Respiratory Tract Infection
Keywords: acute; adaptive cellular immune phenotypes; infants; Lymphocyte; premature; respiratory viral infections
MeSH Terms: conditions — Respiratory Tract Infections; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, blood plasma, blood cells, saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Full-Term Healthy Infants (> /=37 weeks gestational age): 130 male and female term infants born at a gestational age of 37 0/7 to 41 6/7 weeks (Healthy comparator) will be observed for sequential respiratory viral infections, patterns of intestinal and respiratory bacterial colonization, and adaptive cellular immune phenotypes which are associated with increased susceptibility to respiratory infections and long term respiratory morbidity
  Interventions: Device: Respiratory Inductive Plethysmography
- Preterm Infants (<36 weeks gestational age): 150 male and female preterm infants born at gestational age 23 0/7 to 35 6/7 weeks will be observed for sequential respiratory viral infections, patterns of intestinal and respiratory bacterial colonization, and adaptive cellular immune phenotypes which are associated with increased susceptibility to respiratory infections and long term respiratory morbidity
  Interventions: Device: Respiratory Inductive Plethysmography

INTERVENTIONS:
Device: Respiratory Inductive Plethysmography — Respiratory Inductive Plethysmography (RIP) will be used to document thoracoabdominal motion, relative minute ventilation, and apnea during the minimally invasive respiratory assessments (NIRAs). Both Full and Preterm Infants will undergo a respiratory assessment via RIP prior to and after a bronchodilator (albuterol)

SUMMARY:
This clinical study will investigate the relationships between sequential respiratory viral infections, patterns of intestinal and respiratory bacterial colonization, and adaptive cellular immune phenotypes which are associated with increased susceptibility to respiratory infections and long term respiratory morbidity in preterm and full term infants. This is a prospective, cohort study, enrolling at a single center via two sites (URMC and URMC-affiliated Highland Hospital and Rochester General Hospital). Enrollment will be accomplished in approximately 15 - 36 months. The study will enroll 280 subjects, 150 pre-term and 130 full-term.

DETAILED DESCRIPTION:
This clinical study will investigate the relationships between sequential respiratory viral infections, patterns of intestinal and respiratory bacterial colonization, and adaptive cellular immune phenotypes which are associated with increased susceptibility to respiratory infections and long term respiratory morbidity in preterm and full term infants. This is a prospective, cohort study, enrolling at a single center via two sites (URMC and URMC-affiliated Highland Hospital and Rochester General Hospital). Enrollment will be accomplished in approximately 15 - 36 months. The study will enroll 280 subjects, 150 pre-term and 130 full-term. This protocol does not study an agent or intervention. However, the bronchodilator, albuterol, a beta 2 agonist, will be administered as part of the Respiratory Inductive Plethysmography (RIP) pulmonary function assessments. All infants will remain in the study up to 3 years plus 17 weeks, depending on gestational age at birth. The full-term infants are expected to be typically developing newborns and generally healthy. Enrolled newborns will have a sample of cord blood (CB) for evaluation of lymphocyte phenotype and baseline neutralizing antibody titers. Maternal saliva samples will be collected to test exposure to environmental tobacco smoke. A nose, throat and rectal swab will be obtained for the assessment of the respiratory and gut microbiome and testing for known respiratory pathogens and pathogen discovery. Prior to hospital discharge, infants will have an evaluation of lymphocyte phenotype and function, and will undergo a respiratory assessment via RIP prior to and after a bronchodilator. Co-morbidities, familial and environmental risk factors for atopy, asthma and respiratory symptoms will be assessed. Following hospital discharge, all babies (full-term and former preterm infants) will be followed longitudinally through 3 years CGA as outpatients. During the first year of follow-up, all infants will have rectal and nose, throat swabs obtained monthly. Screening for symptomatic respiratory dysfunction and illnesses will also occur during the time of follow-up as per schedule.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Preterm Cohort: - Signed Informed Consent from parent(s) or legal guardian(s) - Preterm infants born at gestational age 23 0/7 to 35 6/7 weeks - Preterm infants admitted to the URMC NICU or Normal Newborn Nursery - Infants less than or equal to 7 days old - Attending physician agreement Inclusion Criteria for Full Term Cohort: - Healthy term infants 37 0/7 to 41 6/7 weeks gestation - Recruited prior to delivery, or from the birthing centers and labor and delivery floor at URMC and Highland Hospital - Infants less than or equal to 7 days old - Signed Informed Consent from parent(s) or legal guardian(s)

Exclusion Criteria:

- Considered to be non-viable (decision made by clinical care team to not provide life-saving therapies) - Known congenital heart disease, not including patent ductus arteriosus (PDA), hemodynamically insignificant ventricular septal defect (VSD) or atrial septal defect (ASD) - Known structural abnormalities of the upper airway, lungs, or chest wall - Known other congenital malformations or syndromes that adversely affect life expectancy or cardiopulmonary development (i.e., neuromuscular disease, trisomy 21) - Known to be born to women who are human immunodeficiency virus (HIV) positive (HIV testing is not required prior to study entry but is available for most mothers-to-be and is performed on all newborns in NY state) - Known congenital or acquired immune deficiency - Family is unlikely to be available for long-term follow-up as determined by the site investigators - No legal guardian who speaks and reads English - Specifically for the term Infants, as healthy infants, they will not have been admitted to the URMC NICU prior to consent. - Any infant with a diagnosis of hypertension, hyperthyroidism, seizures, arrhythmias, or sensitivity to sympathomimetic amines will be excluded from the BDR assessment. - Any infant with hypersensitivity to any of components of albuterol sulfate will be excluded from the BDR assessment. An infant or child with such history may remain eligible for the remainder of the study if they qualify by other inclusion and exclusion criteria.

Ages: 0 Days to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study subjects were enrolled from sequential preterm and full term births at the University of Rochester
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2013-03-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Calculate presence of at/near term gestation cellular immune response to mitogen and antigen specific responses to > /=1 viral pathogens isolated over 1st 2yrs CGA via lymphocyte assessment | 2 years CGA
Degree of adaptive immune system maturation utilizing flow cytometric analysis of lymphocytes in blood | From 41 weeks gestation through 3 years CGA
  Assess blood lymphocyte subsets at birth (cord blood), discharge and at 1 year of age
Degree of immune system maturation utilizing flow cytometric analysis of lymphocytes in umbilical cord blood and peripheral blood | From 41 weeks gestation through 3 years CGA
Etiology of symptomatic viral respiratory infections as assessed by TLDA PCR Assays of biospecimens | 2 years CGA
Number of respiratory tract symptomatic and asymptomatic viral infections weekly. | 41weeks gestation
Number of symptomatic viral respiratory infections | 2 years CGA
Occurrence of respiratory tract viral infections (asymptomatic and symptomatic) | From 37- 41 weeks gestation, through the first 1 and 2 years CGA, respectively
Patterns of respiratory and gut bacterial microbiome as they develop weekly | 41 weeks gestation
Pulmonary function via Respiratory Inductive Plethysmography (RIP) with Bronchodilator Response (BDR) | 41 weeks gestation
Rate of adaptive immune system maturation utilizing flow cytometric analysis of lymphocytes in blood | From 37- 41 weeks, through the first 1 and 3 years CGA
Rate of immune system maturation utilizing flow cytometric analysis of lymphocytes in umbilical cord blood and peripheral blood | 41 weeks gestation
Severity of illness due to viral respiratory tract infections | 2 years CGA
Severity of respiratory tract viral infections (asymptomatic and symptomatic) as assessed by the COAST Respiratory Symptom Scale. | 2 years CGA
Viral load of respiratory pathogens in the nasopharynx of infants with symptomatic RTIs | 2 years CGA

SECONDARY OUTCOMES:
Patterns of respiratory and gut bacterial microbiome as they change monthly from hospital discharge at term or near term gestation | Through the first 1 year CGA
Presence of cord blood antigen-neutralizing antibodies correlates with the presence of specific antigen responses in lymphocytes | At term or near term gestation
Pulmonary function via RIP with BDR | At 1 year CGA and 3 years CGA
Titers of neutralizing antibodies in cord blood to isolated viral pathogens | Through the first 2 years CGA

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center - Strong Memorial Hospital - Infectious Diseases, Rochester, New York, United States

REFERENCES:
- [Result] McDavid A, Corbett AM, Dutra JL, Straw AG, Topham DJ, Pryhuber GS, Caserta MT, Gill SR, Scheible KM, Holden-Wiltse J. Eight practices for data management to enable team data science. J Clin Transl Sci. 2020 Jun 23;5(1):e14. doi: 10.1017/cts.2020.501. PMID 33948240
- [Result] Caserta MT, Yang H, Bandyopadhyay S, Qiu X, Gill SR, Java J, McDavid A, Falsey AR, Topham DJ, Holden-Wiltse J, Scheible K, Pryhuber G. Measuring the Severity of Respiratory Illness in the First 2 Years of Life in Preterm and Term Infants. J Pediatr. 2019 Nov;214:12-19.e3. doi: 10.1016/j.jpeds.2019.06.061. Epub 2019 Jul 31. PMID 31377041

DOCUMENTS (1):
  • Informed Consent Form (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT01789268/ICF_000.pdf